CLINICAL TRIAL: NCT06787235
Title: Nutritional Intervention to Reduce Alcohol Consumption
Acronym: NIRAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-00509
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ketogenic diet (Experimental): The modified Atkins KD is defined as <20g carbohydrate per day with freely allowed protein consumption. Recommended protein and fat intake will be calculated for each participant based on their energy needs.
  Interventions: Dietary Supplement: Modified ketogenic diet
- Nutritional consultation (Active Comparator): Patients in the control group will have the option to receive an individual consultation by a clinical dietician during the inpatient setting, addressing the specific nutritional needs of people with AUD and providing the knowledge of an adequate and balanced diet.
  Interventions: Other: Individual nutritional consultation

INTERVENTIONS:
Dietary Supplement: Modified ketogenic diet — The modified Atkins KD is defined as <20g carbohydrate per day with freely allowed protein consumption. Recommended protein and fat intake will be calculated for each participant based on their energy needs.
  Arms: Modified ketogenic diet
Other: Individual nutritional consultation — The nutritional consultation will be provided by a dietician to improve individual health
  Arms: Nutritional consultation

SUMMARY:
To test whether the implementation of a modified ketogenic diet (KD) is efficient in reducing outcome measures in relation to alcohol consumption in patients with alcohol use disorder (AUD).

DETAILED DESCRIPTION:
This pilot study aims at testing randomization and feasibility of implementing a modified KD in patients with AUD undergoing standard alcohol withdrawal treatment. For this purpose, a a standardized nutritional intervention consisting of interprofessional consultations by clinical dieticians and medical professionals will be implemented. Patients in the control group will be randomized in an AUD as usual treatment with an additional optional nutritional consultation. After dismission of inpatient care, the participants will be followed up for adherence to the modified KD in the outpatient clinic for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* AUD diagnosis according to Diagnostic and Statistical Manual (DSM)-5
* BMI > 22 (because of potential modified KD-side effect of weight loss)
* Able to give informed consent as documented by signature
* Last alcohol drink intake within 72 hours before treatment initiation

Exclusion Criteria:

* Pregnant or lactating women,
* Inability or contraindications to undergo the investigated intervention (BMI<18)
* Clinically significant concomitant diseases impairing reasonable decision making (e.g. psychosis, dementia)
* Inability to follow the procedures of the study, e.g. due to language problems, Previous enrolment in a clinical trial
* Patients undergoing opioid maintenance treatment
* Patients taking medications for drinking relapse prevention
* Patients with a blood hemoglobin A1C (HbA1C) > 7%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Modified ketogenic diet (KD) | 8 weeks
  Patients'adherence to the modified KD during the study by percentage of prospective food intake recording of meal plans and measurement of the state ketosis by capillary blood readings of ketones.

SECONDARY OUTCOMES:
Drinking outcome | 8 weeks
  Phosphatidylethanol level blood measures, Timeline Followback Clinical Interview measured with daily standard drinks of 10 grams of alcohol, Obsessive Compulsive Drinking Scale to assess craving (a 14-item questionnaire that measures an individual's alcohol use and his/her attempts to control his/her drinking, each item scored from 0 to 4)
Nutritional outcome | 8 weeks
  Nutrimental Screener 1.0 - 10 item questionnaire on nutritional habits (bimodal yes/no), Food Frequency 13 item questionnaire on eating habits (5 point Likert scale from never to daily use)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pfeifer, Study Chair — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No